CLINICAL TRIAL: NCT01532245
Title: The Use of Constant-flow Technique for Determining the Lower Inflexion Point of Pressure-volume Curve and Intrinsic PEEP During One-lung Ventilation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DEOEC RKEB/IKEB 3504-2011
Record Dates: First submitted 2012-02-02; First posted 2012-02-14 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: One Lung Ventillation (OLV); Two Lung Ventillation (TLV); Positive End Expiratory Pressure (PEEP); Zero End-expiratory Pressure (ZEEP)
MeSH Terms: interventions — One-Lung Ventilation

ARMS (3):
- two-lung ventilation (TLV) (Active Comparator): During two-lung ventilation (TLV) and OLV 8 ml•kg-1 tidal volume was used.
  Interventions: Other: two lung ventilation (TLV)
- one lung ventillation (OLV) without PEEP (Active Comparator): During OLV, ventilation periods of ten minutes, with and without 5 cmH2O positive end-expiratory pressure (PEEP) were alternated.
  Interventions: Other: one lung ventilation (OLV) without PEEP
- one lung ventilation (OLV) with PEEP (Active Comparator): During OLV, ventilation periods of ten minutes, with and without 5 cmH2Opositive end-expiratory pressure (PEEP) were alternated
  Interventions: Other: One lung ventilation (OLV) with positive end-expiratory pressure (PEEP)

INTERVENTIONS:
Other: two lung ventilation (TLV) — During two-lung ventilation (TLV) and OLV 8 ml•kg-1 tidal volume was used.
  Arms: two-lung ventilation (TLV)
Other: one lung ventilation (OLV) without PEEP — During OLV, ventilation periods of ten minutes, with and without 5 cmH2O positive end-expiratory pressure (PEEP) were alternated.
  Arms: one lung ventillation (OLV) without PEEP
Other: One lung ventilation (OLV) with positive end-expiratory pressure (PEEP) — During OLV, ventilation periods of ten minutes, with and without 5 cmH2O positive end-expiratory pressure (PEEP) were alternated
  Arms: one lung ventilation (OLV) with PEEP

SUMMARY:
One method for treating intraoperative hypoxia during one-lung ventilation (OLV) is application of PEEP to the dependent lung. However, only a minority of patients benefit from this maneuver. The effect of applied PEEP on oxygenation depends on the relation between the total end-expiratory pressure and the lower inflexion point (LIP) of pressure-volume curve (1). LIP during OLV can be determined with super-syringe technique, but is too complicated for routine operating room use. An alternative is the constant-flow method which is easy and widely used in intensive care settings (2). The investigators goal was to confirm that the constant-flow method as applied by an intensive care ventilator works during OLV.

Methods: After IRB approval and written, informed consent, data were obtained from 20 patients during OLV for thoracic surgery who were ventilated with an AVEA (VIASYS Healthcare) critical-care ventilator. During two-lung ventilation (TLV) and OLV 8 ml•kg-1 tidal volume was used. During OLV, ventilation periods of ten minutes, with and without 5 cmH2O PEEP were alternated. During each period, the investigators recorded arterial blood partial pressures, respiratory and hemodynamic values, intrinsic PEEP (PEEPi), and LIP. PEEPi and LIP were determined using the automatic mode of the ventilator; specifically, LIP was determined with a continuous flow of 3L/minute.

ELIGIBILITY:
Inclusion Criteria:

* thoracic surgery lung ventillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
intrinsic positive end-expiratory pressure (PEEP) during ventillation | 10 minutes
  constant-flow method useful for determination of intrinsic positive end-expiratory pressure (PEEPi) during OLV
lower inflexion point (LIP) of P-V curve during one lung ventillation (OLV) | 10 minutes
  constant-low method useful for determination of lower inflexion point (LIP) of P-V curve during one lung ventillation (OLV).
net change of Lower Inflexion Point (LIP)- intrinsic positive end-expiratory pressure (PEEPi) ditstance with PEEP | 10 minutes
  Relationship between the net change of lower inflexion point (LIP)- positive end-expiratory pressure (PEEPi) ditstance with and without positive end-expiratory pressure (PEEP) and change of PaO2 is useful during OLV for determination of patients reaction for application extternal positive end-expiratory pressure (PEEP)
net change of lower inflexion point (LIP)-PEEPi ditstance without PEEP | 10 minutes
  Relationship between the net change of lower inflexion point (LIP)-intrinsic positive end-expiratory pressure (PEEPi) ditstance with and without positive end-expiratory pressure (PEEP) and change of PaO2 is useful during one lung ventillation (OLV) for determination of patients reaction for application external positive end-expiratory pressure (PEEP).

CONTACTS AND LOCATIONS:
Overall Officials: Tamás Végh,, M.D., Principal Investigator — Klinikum Ludwigshafen